CLINICAL TRIAL: NCT00661648
Title: Prevention for Surgical Site Infection After Pancreatic Resection
Brief Title: Effect of an Artificial Pancreas in Patients Undergoing Pancreatic Resection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kochi University (Other)
Responsible Party: Kochi University, Kochi Medical School
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TGC-AP-03; Kochi University
Record Dates: First submitted 2008-04-14; First posted 2008-04-18 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Pancreatic Diseases
Keywords: surgery
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): glucose levels were controlled using sliding scale
- 2 (Experimental): received programmed infusions of insulin determined by the control algorithm of the artificial pancreas
  Interventions: Device: the closed-loop STG-22 system (Nikkiso Inc, Tokyo, Japan)

INTERVENTIONS:
Device: the closed-loop STG-22 system (Nikkiso Inc, Tokyo, Japan) — artificial pancreas
  Other Names: an artificial pancreas system (Nikkiso Inc, Tokyo, Japan)
  Arms: 2

SUMMARY:
This study evaluated that strict control of perioperative blood glucose following pancreatic resection by using an artificial pancreas would improve postoperative surgical site infection.

DETAILED DESCRIPTION:
This study recruited 50 patients undergoing elective pancreatic resection for pancreatic diseases. Perioperative blood glucose concentration was continuously monitored using an artificial pancreas system. We prospectively divided into two groups: one for whom glucose levels were controlled using a manual injection of insulin according to the commonly used sliding scale and another that received programmed infusion of insulin determined by the control algorithm of the artificial pancreas.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective pancreatic resection for pancreatic diseases.

Exclusion Criteria:

* weight loss greater than 10% during the previous 6 months
* sign of distant metastasis
* respiratory, renal, or heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
the incidence of surgical site infection | 30th postoperative day

SECONDARY OUTCOMES:
the incidence of hypoglycemia and cost during the hospitalization | during the hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Takehiro Okabayashi, MD, Study Director — Kochi Medical School
Locations (1):
- Kochi Medical School, Nankoku, Kochi, Japan